CLINICAL TRIAL: NCT07114302
Title: Effects of Digitally-Assisted Brief Behavioral Treatment for Insomnia in College Students: A Randomized Controlled Trial
Brief Title: Digitally-Assisted Brief Behavioral Treatment for Insomnia in College Students
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Hsiao-Yean Chiu, Principal Investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N202502044
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Insomnia
Keywords: college students; Digitally-Assisted BBTI; BBTI; undergrate students
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- interactive e-book BBTI group (Experimental): Participants will experience 5-week treatment period (1 in person and 4 via message).
  Interventions: Behavioral: Interactive E-book BBTI Group
- BBTI-APP group (Experimental): Participants will experience 5-week treatment period (1 in person and 4 via message).
  Interventions: Behavioral: BBTI-APP Group
- sleep hygiene group (No Intervention): Participants will received sleep hygiene at the enrollment of the study and be required to maintain their usual lifestyle and medical treatment for 5 weeks.

INTERVENTIONS:
Behavioral: Interactive E-book BBTI Group — Researchers will guide you on how to use the interactive e-book and help install it on your smartphone. Over the next four weeks, you will be asked to record your sleep diary daily. You will use the e-book to perform sleep stimulus control, sleep restriction, and relaxation techniques to promote better sleep. Researchers will contact you via LINE during the second and fourth weeks, and may call you if necessary.
  Arms: interactive e-book BBTI group
Behavioral: BBTI-APP Group — Researchers will assist you in creating an account for the mobile application and will explain the interface and how to operate it. Over the next four weeks, you will be asked to record your sleep diary daily. You will use the mobile app to carry out sleep stimulus control, sleep restriction, and relaxation techniques to improve sleep. Researchers will contact you via LINE during the second and fourth weeks, and may call you if necessary.
  Arms: BBTI-APP group

SUMMARY:
The study is a single-blind study, parallel randomized controlled trial method. The purpose of this study was to explore the effectiveness of the mobile version of Application based Brief Behavioral Treatment for Insomnia (BBTI-APP) and the interactive e-book version of BBTI in improving the severity of insomnia, sleep quality and mood among college students. Measurement outcomes are sleep parameters measured by the Chinese version of Insomnia Severity Index, Chinese version of The Depression, Anxiety and Stress Scale - 21 Items, and sleep diary. Questionnaires will be assessed in pretreatment, posttreatment, and one-month follow-up. We hypothesized that compared with the sleep hygiene group, both the BBTI-APP and the interactive e-book BBTI can significantly improve college students' insomnia symptoms, emotional distress, and quality of life.

DETAILED DESCRIPTION:
Background： Insomnia is a common health problem faced by college students. It not only causes poor academic performance and reduces the quality of life, but also increases the risk of mood disorders and suicide. However, insomnia among college students has long been ignored by health care providers. Currently, insomnia drugs and cognitive behavioral therapy for insomnia are mostly used clinically to treat insomnia. However, there are no long-term use guidelines for insomnia drugs for teenagers. Cognitive behavioral therapy for insomnia is a treatment that is expensive, time-consuming, and lacks accessibility.

Purpose： The purpose of this study was to explore the effectiveness of the mobile version of Application based Brief Behavioral Treatment for Insomnia (BBTI-APP) and the interactive e-book version of BBTI in improving the severity of insomnia, sleep quality and mood among college students. We hypothesized that compared with the sleep hygiene group, both the BBTI-APP and the interactive e-book BBTI can significantly improve college students' insomnia symptoms, emotional distress, and quality of life.

Method： The study is a single-blind study, parallel randomized controlled trial method. It is anticipate to include 30 college students, who will be randomly assigned to the BBTI-APP group (10 people) and the interactive e-book BBTI group (10 people) in a ratio of 1:1:1. and sleep hygiene team (10 people). If assigned to the BBTI-APP group, college students can use the mobile phone app to record sleep, watch BBTI treatment content and sleep hygiene, perform muscle relaxation and listen to relaxing music. The study intervention time is four weeks in total.

Anticipated Results：

1. BBTI-APP and interactive e-book BBTI can effectively improve the severity of insomnia, sleep quality and mood of college students
2. It enables researchers to gain relevant knowledge and experience in using BBTI-APP and BBTI e-books to improve college students' insomnia severity, sleep quality and mood.

Keywords：Digital, Brief Behavioral Treatment for Insomnia,BBT-I, insomnia, mood, college students

ELIGIBILITY:
Inclusion Criteria: With an electronic mobile device that can access the Internet, reporting insomnia including falling asleep more than three days a week or being awake at night for ≥30 minutes for more than 3 months, screened by the Chinese version of the Insomnia Severity Index- Chinese Version -C, with a total score of ≥10 points, can communicate in Chinese and complete the research questionnaire -

Exclusion Criteria: Those entering internship, shift workers, those with a history of epilepsy, those with other sleep disorders such as sleep apnea, those currently diagnosed with mental illness, substance abuse or alcohol addiction.

-

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Sleep parameters from sleep logs: sleep onset latency(SOL) | At baseline, week 1 to 4 (during the intervention), and one month (follow-up)
  Sleep onset latency(SOL) is the time of duration from lying on bed to fall asleep. SOL shorter than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: after sleep onset(WASO) | At baseline, week 1 to 4 (during the intervention), and one month (follow-up)
  Wake after sleep onset(WASO) is the total time of wakefulness after sleep onset. WASO less than 30 minutes is one of criteria of good sleep condition.
Changes in Sleep parameters from sleep logs: total sleep time(TST) | At baseline, week 1 to 4 (during the intervention), and one month (follow-up)
  Total sleep time(TST) is the total time of falling asleep. TST will be used to calculate sleep efficiency(SE).
Changes in Sleep parameters from sleep logs: sleep efficiency(SE) | Time Frame: At baseline, week 1 to 4 (during the intervention), and one month (follow-up)
  Sleep efficiency(SE) is the percentage of total sleep time to time in bed. A good sleep condition should meet the criteria of SE greater than 85%.
Changes in Insomnia Severity | At baseline, week 5 (after the intervention), and one month (follow-up)
  Insomnia Severity will be measured by Chinese version Insomnia Severity Index (ISI). ISI has 7 questions to evaluate sleep difficulty. The total score range from 0-28, if score>7 is associated with insomnia. The higher score means more severe insomnia.

SECONDARY OUTCOMES:
Changes in Depression | At baseline, week 4 (after the intervention), and one month (follow-up)
  Depression will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of depression.
Changes in Anxiety | At baseline, week 4 (after the intervention), and one month (follow-up)
  Anxiety will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of anxiety. The total score should be multiplied by 2 range from 0-42, if score>7 is associated with anxiety. The higher score means more severe anxiety.
Changes in Stress | At baseline, week 4 (after the intervention), and one month (follow-up)
  Stress will be measured by Depression Anxiety Stress Scale-21 (DASS21). DASS21 has 21 questions to evaluate the state of depression, anxiety, and stress. 7 of the questions are used to measure the severity of stress. The total score should be multiplied by 2 range from 0-42, if score>14 is associated with anxiety. The higher score means more severe stress.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Medical University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No